CLINICAL TRIAL: NCT07158086
Title: Molecular Underpinnings of Heart Failure, Integrative Multi-Omics, and Non-Coding RNA Profiling: the BIOCARDIUM-HF Study
Brief Title: Molecular Underpinnings of Heart Failure, Integrative Multi-Omics, and Non-Coding RNA Profiling
Acronym: BIOCARDIUM-HF
Status: Not yet recruiting | Type: Observational
Sponsor: University of Zurich (Other)
Responsible Party: Principal Investigator, Jan Kleeberger, Principal Investigator, University of Zurich
Other Study IDs: 25_0908
Record Dates: First submitted 2025-08-27; First posted 2025-09-05 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Heart Failure; Heart Failure (for Example, Fluid Overload)
MeSH Terms: conditions — Heart Failure; Edema

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Heart Failure with reduced ejection fraction (HFrEF): LVEF <40%
- Heart Failure with preserved ejection fraction (HFpEF): LVEF >50%
- Heart Failure with mildyly reduced ejection fraction (HFmrEF): LVEF >40% and <50%

SUMMARY:
The main objective of the study is to achieve a comprehensive phenotyping of patients with heart failure, combining detailed clinical characterization with in-depth molecular profiling. By integrating clinical data with cutting-edge multi-omics techniques (including transcriptomics, epigenomics, and proteomics), this research aims to identify molecular signatures, particularly non-coding RNAs (ncRNAs), that are linked to the onset and progression of HF. Through advanced molecular profiling of biological samples and the analysis of clinical parameters, including advanced imaging, hemodynamic profiling, and biomarker analysis, the study will contribute to the deep phenotyping of HF patients.

The secondary objective aims to uncover potential biomarkers that may serve as predictive indicators of disease progression and identify novel therapeutic targets, offering promising avenues for future treatments in this challenging patient population.

ELIGIBILITY:
INCLUSION CRITERIA

* Female and Male, age ≥18 years at screening.
* Diagnosis of Heart Failure according to ESC Heart Failure Guidelines
* Ability to understand the requirements of the study and to provide informed consent.
* Willingness to undergo follow-up.

EXCLUSION CRITERIA

Patients will be excluded if they meet any of the following conditions:

* Active malignancy or history of cancer with ongoing treatment (e.g., chemotherapy, radiotherapy, immunotherapy).
* Autoimmune or systemic inflammatory diseases.
* Concomitant infections, including acute systemic infections (e.g., sepsis, pneumonia) or chronic infections with systemic impact (e.g., HIV, hepatitis B/C with elevated transaminases).

Other exclusion criteria:

* Age<18 years old
* Inability to provide written informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study aims to enroll all patients presenting with clinical signs and symptoms of acute heart failure. As this is an all-comer cohort, the investigators expect no selection bias in terms of sex and gender.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2030-11-30 (Estimated); Study Completion 2031-11-30 (Estimated)

PRIMARY OUTCOMES:
Death from any cause | From enrollment up to five years
Heart failure hospitalization | From enrollment up to five years

CONTACTS AND LOCATIONS:
Overall Officials: Jan A Kleeberger, MD, Principal Investigator — Universitätsspital Zürich; Francesco Paneni, MD, PhD, Study Director — University of Zurich
Locations (1):
- University Hospital of Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided